CLINICAL TRIAL: NCT02279524
Title: A Phase IIb, Double Blind Randomized, Controlled Clinical Trial, to Evaluate the Efficacy and Safety of Two Aramchol Doses Versus Placebo in Patients With Non-Alcoholic Steatohepatitis (NASH) - Aramchol 005 Study
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Two Aramchol Doses Versus Placebo in Patients With NASH
Acronym: Aramchol_005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galmed Research and Development, Ltd. (Industry)
Collaborators: Sharp (Industry); Diamond Pharma Services Regulatory Affairs Consultancy (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); ClinIntel (Industry); Itamar-Medical, Israel (Industry); One Way Liver OWL (Industry); Medical University of Graz (Other); Tel-Aviv Sourasky Medical Center (Other Government); DSG EDC (Unknown); TransPerfect (Industry); Clinical Reference Laboratory (Industry)
Responsible Party: Sponsor
Organization: Galmed Pharmaceuticals Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aramchol005
Record Dates: First submitted 2014-10-23; First posted 2014-10-31 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Fatty Liver; Non-Alcoholic Steatohepatitis; Liver Diseases; Liver Fibroses
Keywords: NASH; fibroses; obesity; diabetes
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Liver Diseases; Liver Cirrhosis; Fibrosis; Obesity; Diabetes Mellitus | interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aramchol 600mg (Experimental): One tablet of Aramchol 400 mg and one tablet of Aramchol 200 mg.
  Interventions: Drug: Aramchol
- Aramchol 400mg (Experimental): One tablet of Aramchol 400 mg and one tablet of matching placebo for Aramchol.
  Interventions: Drug: Aramchol
- Placebo (Placebo Comparator): Two tablet of Aramchol matching placebo.
  Interventions: Drug: Aramchol

INTERVENTIONS:
Drug: Aramchol — Subjects will be administered Aramchol as follows:
  * One tablet of Aramchol 400 mg and one tablet of matching placebo for Aramchol.
  * One tablet of Aramchol 400 mg and one tablet of Aramchol 200 mg.
  * Two tablet of Aramchol matching placebo. The tablets should be taken orally in the morning within 30 min after breakfast with a glass of water (250 ml).
  Subjects are allowed to omit study drugs up to 3 consecutive days during the study.
  Other Names: Placebo

SUMMARY:
This is a multicenter, Phase IIb, randomized, double blind, placebo-controlled study designed to evaluate the efficacy and safety of two Aramchol doses in subjects that are 18 to 75 years of age, with Non-Alcoholic Steatohepatitis (NASH) confirmed by liver biopsy performed in a period of 6 months before entering the study, with overweight or obesity and who are pre diabetic or type II diabetic.

Eligible subjects will be enrolled into three treatments arms: Aramchol 400 and 600 mg tablets and placebo tablets in ratio 2:2:1.

The subjects will be evaluated at study sites for 11 scheduled visits during one year (52 weeks). After completion of the study treatment period, the subjects will be followed for an additional period of 13 weeks without study medication (until visit 11 (week 65)).

DETAILED DESCRIPTION:
This is a multicenter, Phase IIb, randomized, double blind, placebo-controlled study designed to evaluate the efficacy and safety of two Aramchol doses in subjects that are 18 to 75 years of age, with Non-Alcoholic Steatohepatitis (NASH) confirmed by liver biopsy performed in a period of 6 months before entering the study, with overweight or obesity and who are pre diabetic or type II diabetic.

Eligible subjects will be enrolled into three treatments arms: Aramchol 400 and 600 mg tablets and placebo tablets in ratio 2:2:1.

The subjects will be evaluated at study sites for 11 scheduled visits: at screening (visit 1(weeks -4 - 0)), baseline (visit 2 (day 0)), visit 3 (week 2), visit 4 week 4), visit 5 (week 8), visit 6 (week 12), visit 7 (week 24), visit 8 (week 32), visit 9 (week 40) and visit 10 (week 52 - (End of Treatment/early termination visit)). After completion of the study treatment period, the subjects will be followed for an additional period of 13 weeks without study medication (until visit 11 (week 65)).

During the screening period, the severity of the disease will be evaluated with blood tests, liver biopsy and NMRS.

During the study the following assessments will be performed:

* Vital signs will be measured at each study visit.
* A physical examination will be performed at the screening visit, 24 weeks, End of Treatment/early termination and week 65 visit.

The following blood tests will be performed: complete blood count (CBC), serum chemistry (including electrolytes, liver enzymes, direct and total bilirubin, glucose, lipid profile which include triglyceride, cholesterol, HDL, LDL and VLDL, CPK, creatinine, urea, albumin, alkaline phosphatase), ESR and urinalysis during the screening visit, baseline, week 2, 4, 8, 24, 40, 52 and 65 (end of follow up) visits. Serology (HBV, HCV and HIV) will be performed during the screening visit. Coagulation (fibrinogen, PT/INR, aPTT) will be measured during screening and at baseline, week 24, End of Treatment/early termination and week 65 visits. Insulin (HOMA) will be measured during the screening, at week 24 and End of Treatment/early termination visits. HbA1C will be measured during the screening, at week 8, 24, 40 and End of Treatment/early termination visits. C reactive protein, Leptin and Adiponectin will be measured during baseline visit and at end of treatment period. The blood samples taken at these visits, will be tested for possible biomarkers. TSH, T3 and T4 will be measured during the screening visit. beta-hCG in women of childbearing potential will be performed during the screening visit. A serum sample will be collected and kept frozen until study end in case special investigation needs to be performed. This sample will be collected during the screening and visit 10/Early Termination.

* Body weight and waist circumference will be measured in screening, baseline, week 24, end of treatment and week 65 visits. Height will be measured during the screening visit.
* ECG will be performed during the screening visit, visit 7 (week 24) and end of treatment visits.
* All subjects will undergo two NMRS scans, at screening and end of treatment visits.
* FibroMax test will be performed only if the investigator thinks it is necessary
* Liver biopsy will be conducted during the screening and end of treatment visit. The biopsy in the screening visit will be performed only if it was not done within the 6 months prior to this visit.
* Metabolomics blood test will be performed at the screening, visit 7 and the End-of-Treatment/Early Termination visits. From some consenting patients (about 15) a sample from the liver biopsy will be taken for analysis.
* Endothelial Function will be conducted in selected sites. The test will be conducted during the baseline visit before the study treatment will be given and End of Treatment/early termination visit.
* Blood sample for Aramchol trough level will be collected (pre-dose) from patients in Israel at baseline (visit 2) week 4 (visit 4), week 12 (visit 6), week 24 (visit 7), week 40 (visit 9), end of treatment (visit 10) and follow up (visit 11). At selected sites in Mexico, USA and Hong Kong one blood sample will be collected (pre-dose) on visit 4 (up to 10 subjects per country) to test for trough Aramchol blood level differences between populations (e.g., African American, Asian, Hispanic).
* Blood sample for gene analysis will be taken from all consenting patients during the baseline visit, will be kept frozen and analyzed only at the study end.
* Life style questionnaire will be completed at all visits.
* Adverse events will be monitored throughout the study.
* Concomitant Medications will be monitored throughout the study.
* Telephone contacts will be performed on week 16, 20, 28, 36, 44 and 48. An interim safety analysis will be conducted as soon as 120 subjects will completed the follow up period of 24 weeks under study treatment. An independent DSMB will analyze the safety data and recommend a continued course of action. All patients will continue to be treated under the study protocol until conclusion of the analysis will be known.

Safety assessment will include frequency and severity of treatment-emergent AEs, clinically significant laboratory abnormalities, ECG changes and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 to 75 years.
2. BMI between 25kg/m2 to 40kg/m2 or waist circumference between 88 cm to 200 cm for women, and between 102 cm to 200 cm for men. If there is deviation above the upper limit, please consult the MRI center, to ensure that the machine is suitable for the patient.
3. Known type II Diabetes Mellitus or pre-Diabetes according to American Diabetes Association. One of the following 3 criteria is needed for pre-Diabetes: Fasting Plasma Glucose > 100mg/dl (5.5 mmol/l) or 2hPG following 75g OGTT > 140 (7.8 mmol/l) mg/dl or HbA1c > 5.7%. HbA1c can be repeated at Investigator's discretion.
4. Histologically proven Steatohepatitis on a diagnostic liver biopsy performed either during screening or within 6 months before screening visit, confirmed by central laboratory reading of the slides.(Steatosis ≥1 + inflammation ≥1 + ballooning ≥1).Total activity NAS score of 4 or more.
5. Liver fat concentration in the liver of 5.5% or more as measured by NMRS.
6. Biopsies with an activity NAS score of 4 or more.
7. Normal synthetic liver function (serum albumin >3.2g/dl, INR 0.8-1.2, conjugated bilirubin < 35 µmol/L).
8. Understanding the nature of the study and signature of the written informed consent.
9. Negative pregnancy test at study entry for females of child bearing potential.
10. Females of child bearing potential practicing reliable contraception throughout the study period (including oral contraceptives) as well as negative pregnancy test at study entry.
11. Hypertensive patients must be well controlled by stable dose of anti-hypertensive medication for at least 2 months prior to screening.
12. Patients previously treated with vitamin E (>400IU/day), Polyunsaturated fatty acid (>2g/day) or Ursodeoxycholic acid or fish oil can be included if stopped or at least maintained on stable dose at least 3 months prior to diagnostic liver biopsy (and are not started during the trial). These treatments-dosages are allowed if they were stable for at least 12 months prior to biopsy and can remain stable throughout the study. (Dosages less than the amounts stated above are allowed without washout- or stable-period restrictions).
13. For patients with type II Diabetes, glycaemia must be controlled (Glycosylated Hemoglobin A1c ≤9%) while any HbA1c change should not exceed 1.5% during 6 months prior to enrolment). Treatments with anti-diabetic medications (except for those mentioned in Exclusion 16) are permitted if glycaemia is self-monitored by the patient. HbA1c can be repeated at Investigator's discretion.

Exclusion Criteria:

1. Patients with other active (acute or chronic) liver disease other than NASH (e.g. viral hepatitis, unless eradicated at least 3 years prior to screening; genetic hemochromatosis; Wilson disease; alpha 1antitripsin deficiency; alcohol liver disease; drug-induced liver disease) at the time of randomization.
2. Patients with clinically or histologically documented liver cirrhosis
3. Known alcohol and/or any other drug abuse or dependence in the last five years.
4. Known history or presence of clinically significant cardiovascular, gastrointestinal, metabolic other than Diabetes Mellitus, neurologic, pulmonary, endocrine, psychiatric, neoplastic disorder or nephrotic syndrome, that in the opinion of the Investigator warrant exclusion from the study.
5. Patients with familial (i.e., genetic) hypertriglyceridemia and familial (i.e., genetic) hypercholesterolemia.
6. History or presence of any disease or condition known to interfere with the absorption distribution, metabolism or excretion of drugs including bile salt metabolites (e.g. inflammatory bowel disease (IBD)), previous intestinal (ileal or colonic) operation, chronic pancreatitis, celiac disease or previous vagotomy. Ongoing Chronic constipation
7. Patients with heart or brain pacemaker (i.e., implantable neurological devices).
8. Surgery during the last three month before screening which involved stent implantation of metal devices (e.g. knee, hip etc.)
9. Weight loss of more than 5% within 6 months prior to randomization.
10. History of bariatric surgery within 5 years of liver biopsy.
11. Uncontrolled arterial hypertension.
12. Women who are pregnant and breast feeding.
13. Diabetes Mellitus other than type II (type I, endocrinopathy, genetic syndromes etc.).
14. Patients with HIV infection.
15. Daily alcohol intake >20 g/day for women and >30 g/day for men (on average per day) as per medical history.
16. Treatment with other anti-diabetic medications:

    GLP-1 receptor agonists and Thiazolidinediones (TZDs), unless started at least 12 months prior to biopsy and on stable dose for 6 months. In case of GLP-1 receptor agonists stopped, it should be at least 6 months before biopsy as per medical history.
17. SGLT-2 Inhibitors, Metformin, fibrates, statins, insulin, DPP-4 inhibitors and sulfonylurea unless prescribed dose has been stable for the last 6 months prior to the biopsy.
18. Treatment with Valproic acid, Tamoxifen, Methotrexate, Amiodarone or chronic treatment with anti-cholinergic agents, corticosteroids, high dose estrogen and tetracycline within 12 months prior to the screening visit.
19. Chronic treatment with antibiotics (e.g. Rifaximin).
20. Homeopathic and/or alternative treatments. Any treatment should be stopped during the screening period at least 48 hours before randomization.
21. Uncontrolled hypothyroidism defined as Thyroid Stimulating hormone >2X the upper limit of normal (ULN). Thyroid dysfunction controlled for at least 6 months prior to screening is permitted.
22. Patients with renal dysfunction eGFR< 40.
23. Unexplained serum creatine phosphokinase (CPK) >3X the upper limit of normal (UNL). Patients with a reason for CPK elevation may have the measurement repeated prior to randomization; a CPK retest > 3X ULN leads to exclusion.
24. Patients with condition(s) that makes them unsuitable to perform the NMRS (as determined by the PI or the MRI facility).
25. Hypersensitivity to Aramchol or to any of the excipients in the tablets
26. Hypersensitivity to cholic acid or bile acid sequestrants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Ratziu, MD, PhD, Principal Investigator — Professor of Hepatology, Université Pierre et Marie Curie & Hospital Pitie Salpetriere Medical University, Paris.
Locations (77):
- United States (17):
  - Profil Institue for Clinical Research Inc., Chula Vista, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empoire Liver Foundation, Rialto, California
  - University of California Department of Medicine Division of Gastroenterology, San Diego, California
  - Orange County Research Center, Tustin, California
  - Indiana University, Indianapolis, Indiana
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research, Raleigh, North Carolina
  - Texas Digestive Disease Consultants, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Gastroenterology Consultants of San Antonio, Live Oak, Texas
  - Texas Liver Institute San Antonio, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- Chile (5):
  - Biomedica Research Group, Santiago
  - Centro de Investigacion Clinica CEIC, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar
- France (8):
  - Centre Hospitalier Universitaire (CHU) d'Angers, Angers
  - Centre Hospitalier Universitaire Dijon Bourgogne, Dijon
  - San Joseph Service Hepato Gastro Entrologie, Marseille
  - Hospital Saint Eloi, Montpellier
  - CHU Centre Hospiatalier Universitaire de Rennes, Paris
  - Hospital Pitie-Salpetriere, Paris
  - Hospital Saint-Antoine AP-HP, Paris
  - Hopital Paul Brousse, Villejuif
- Georgia (5):
  - Unimed Adjara, Batumi
  - Clinic Cortex, Tbilisi
  - David Tatishvili Medical Center, Tbilisi
  - LTD Diacor, Tbilisi
  - Research Institute of Clinical Medicine, Tbilisi
- Germany (3):
  - Medizinische Hochschule, Hanover
  - EUGASTRO GmbH, Leipzig
  - Universitat Leipzig Medizinische Fakultat, Leipzig
- Humanity & Health Medical Centre, Central, Hong Kong
- Israel (8):
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Ein Karem Medical Cente, Jerusalem
  - Naharia Medical Center, Nahariya
  - The Holy family Medical Center, Nazareth
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Saurasky Medical Center, Tel Aviv
  - Asaf Harofeh Medical Center, Zrifin
- Italy (13):
  - Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O. San Paolo, Milan
  - A.O. U. "Federico II" di Napoli, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale "A.Cardarelli", Napoli
  - Azienda Ospidaliera Universitaria Seconda Universita di Napoli, Napoli
  - A.O.U. Maggiore della Carità, Novara
  - "Ospedale Cristo Re" dell'Istituto Figlie di N.S. al Monte Calvario, Roma
  - Fondazione Policlinico di Tor Vergata, Roma
  - Ospedale San Camillo, Roma
  - Policlinico A. Gemelli, Roma
  - Policlinico Umberto I Di Roma, Roma
  - Policlinico Univestitario Campus Biomedico, Roma
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vilinius University Hospital Santariskiu Klinikos, Vilnius
- Mexico (9):
  - Unidad de Hígado Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León
  - JM Research, Cuernavaca
  - Consultorio Médico, Metepec
  - Torre de Consultorios Clinica Londres, Mexico City
  - Consultorio Medico del Dr. Mauricio Castillo Barradas, Mexico City
  - Consultorio Medico, Mexico City
  - Instituto de Ciencias Medicas y de la Nutricion Salvador Zubiran, Mexico City
  - Accelerium Clinical Research, Monterrey
  - "Angeles Valle oriente" Hospital, San Pedro Garza García
- Romania (5):
  - Clinical Institute Colentina, Bucharest
  - The National Institute for Infectious Diseases "Prof. Dr. Matei Bals", Clinical Department for Adults II, Bucharest
  - Cluj County Emergency Hospital, Cluj-Napoca
  - TVM Medical, Cluj-Napoca
  - County Hospital Mures-Gastroenterology Department, Târgu Mureş

REFERENCES:
- [Derived] Ratziu V, de Guevara L, Safadi R, Poordad F, Fuster F, Flores-Figueroa J, Arrese M, Fracanzani AL, Ben Bashat D, Lackner K, Gorfine T, Kadosh S, Oren R, Halperin M, Hayardeny L, Loomba R, Friedman S; ARREST investigator study group; Sanyal AJ. Aramchol in patients with nonalcoholic steatohepatitis: a randomized, double-blind, placebo-controlled phase 2b trial. Nat Med. 2021 Oct;27(10):1825-1835. doi: 10.1038/s41591-021-01495-3. Epub 2021 Oct 7. PMID 34621052

RESULTS

PARTICIPANT FLOW:
Groups:
- Aramchol 600mg: One tablet of Aramchol 400 mg and one tablet of Aramchol 200 mg, once a day for 52 weeks
- Aramchol 400mg: One tablet of Aramchol 400 mg and one tablet of matching placebo for Aramchol, once a day for 52 weeks
- Placebo: Two tablets of matching placebo for Aramchol, once a day for 52 weeks
Period: Overall Study
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Started | 98 | 101 | 48
Completed | 88 | 90 | 41
Not Completed | 10 | 11 | 7
Not completed — Withdrawal by Subject | 3 | 6 | 3
Not completed — Adverse Event | 4 | 3 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Disallowed medication | 1 | 1 | 2
Not completed — Bariatric surgery | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo | Total
Number analyzed (Participants) | 98 | 101 | 48 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (9.8) | 53.9 (10.9) | 54.4 (10.3) | 54.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 65 | 25 | 160
  Male | 28 | 36 | 23 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 4 | 1 | 10
  Black or African American | 1 | 0 | 1 | 2
  Hispanic | 12 | 17 | 11 | 40
  Latin | 16 | 14 | 3 | 33
  Latin American | 1 | 1 | 1 | 3
  Latin Race | 0 | 1 | 1 | 2
  Mixed (Martinican) | 0 | 1 | 0 | 1
  White | 63 | 63 | 30 | 156
BMI (kg/m^2) at Screening [Mean (Standard Deviation); unit: kg/m^2] | 33 (4.2) | 32.4 (4.5) | 32.6 (4.9) | 32.7 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Liver Fat
Description: absolute % change from baseline to end of study in liver triglycerides to water ratio (fat/water+fat) as measured by MRS
Time Frame: At screening (baseline) and at week 52
Population: Pre-defined FASmri analysis set
Measure: Mean (Standard Deviation); unit: Abs. % Change from Baseline Liver Fat
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 83 | 90 | 41
Abs. % Change from Baseline Liver Fat | -3.18 (1.01) | -3.41 (0.96) | -0.09 (1.38)
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.0655, Mixed Models Analysis; Difference in least square means = -3.09; Post-Hoc Responder Analysis - was also carried out. See Post-Hoc analysis
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.0450, Mixed Models Analysis; Difference in least square means = -3.32; Post-Hoc Responder Analysis - was also carried out. See Post-Hoc analysis

2. Secondary Outcome: NASH Resolution Without Worsening of Fibrosis
Description: The endpoint was defined as end of study biopsy, observed under microscope and showing:
  * Cell Ballooning (special form of liver cell injury associated with cell swelling and enlargement)= 0
  * Inflammation (presence or absence of cells from the immune system) = 0 or 1
  * No worsening of fibrosis (scar formation) = increase in fibrosis score by 1 or more point
Time Frame: At screening and at week 52
Population: FASBiopsy analysis set
Measure: Number; unit: % of subjects reaching the end-point
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 78 | 80 | 40
% of subjects reaching the end-point | 16.7 | 7.5 | 5
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.0514, Regression, Logistic; The method used was a Baseline Adjusted Logistic Regression; Odds Ratio (OR) = 4.74, 95% CI 2-sided [0.99 to 22.66]
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.4955, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.33 to 9.61]

3. Secondary Outcome: Fibrosis Improvement Without Worsening of NASH
Description: The endpoint was defined as end of study biopsy showing:
  * A decrease in fibrosis score ≥ 1 point
  * No worsening of NASH (defined by an increase of inflammation and/or ballooning)
Time Frame: At screening and at week 52
Population: Predefined FASBiopsy analysis set
Measure: Number; unit: % of subjects reaching the end-point
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 78 | 80 | 40
% of subjects reaching the end-point | 29.5 | 21.3 | 17.5
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.2110, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.70 to 5.04]
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.8425, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.40 to 3.05]

4. Secondary Outcome: Change From Baseline to Week 52/Termination in ALT
Description: Change from baseline to Week 52 or Termination visit in ALT levels (U/L)
Time Frame: At baseline until week 52
Population: Pre-defined FASALT analysis set
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 98 | 100 | 47
U/L | -17.3 (3.7) | -12.0 (3.6) | 11.8 (5.2)
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least square means = -29.1, Standard Error of Mean 6.4
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Difference in least square means = -23.8, Standard Error of Mean 6.3

5. Other Pre Specified Outcome: Change From Baseline to Termination/Early Termination in HbA1C
Description: Change from baseline to Week 52 or Termination visit in Hemoglobin A1C (%)
Time Frame: At baseline until week 52
Population: Analysis Set: FASHgA1C
Measure: Least Squares Mean (Standard Error); unit: % of HbA1C
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 96 | 98 | 47
% of HbA1C | -0.1268 (0.0769) | -0.0417 (0.0754) | 0.3202 (0.1089)
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Difference in least square means = -0.4470, 95% CI 2-sided [-0.7063 to -0.1877]
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.0061, Mixed Models Analysis; Difference in least square means = -0.3620, 95% CI 2-sided [-0.6196 to -0.1043]

6. Post Hoc Outcome: Change From Baseline to Week 52/Termination in AST
Description: Change from baseline to Week 52 or termination visit in AST levels (U/L)
Time Frame: At baseline until week 52
Population: FASAST Analysis Set
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 98 | 100 | 47
U/L | -10.83 (2.49) | -7.21 (2.42) | 6.68 (3.50)
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least square means = -17.5, Standard Error of Mean 4.2
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.0011, Mixed Models Analysis; Difference in least square means = -13.9, Standard Error of Mean 4.2

7. Post Hoc Outcome: Change From Baseline in Mean Liver Fat - Responder Analysis
Description: A responder is defined according to >5% absolute improvement from baseline. A cutoff of 5% absolute reduction in liver F/(F+W) ratio was used as a surrogate for potentially clinically meaningful MRI reduction.
Time Frame: Baseline to 52 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 83 | 90 | 41
percentage of participants | 47.0 | 36.7 | 24.4
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.0279, Mixed Models Analysis; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.11 to 6.88]
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.0878, Regression, Logistic; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.89 to 5.46]

8. Post Hoc Outcome: Progression to Cirrhosis
Description: Fibrosis stage 4 in liver biopsy
Time Frame: Week 52
Population: This analysis is limited by low number of events, and the duration of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
Number analyzed (Participants) | 78 | 80 | 40
Participants | 1 | 6 | 3
Statistical Analysis 1: Comparison: Aramchol 600mg vs Placebo; Test type: Superiority; p = 0.1008, Regression, Logistic; Odds Ratio (OR) = 0.14, 95% CI 2-sided [0.01 to 1.46] — This analysis is limited by low number of events, and the duration of the study
Statistical Analysis 2: Comparison: Aramchol 400mg vs Placebo; Test type: Superiority; p = 0.5693, Regression, Logistic; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.13 to 3.05] — This analysis is limited by low number of events, and the duration of the study

ADVERSE EVENTS:
Time Frame: 52 weeks + 13 weeks follow-up
Arm/Group | Aramchol 600mg | Aramchol 400mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/101 | 0/48
Serious Adverse Events (participants affected / at risk) | 9/98 | 9/101 | 6/48
Other Adverse Events (participants affected / at risk) | 77/98 | 75/101 | 33/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aramchol 600mg (N=98) | Aramchol 400mg (N=101) | Placebo (N=48)
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Mammogram abnorma (Investigations) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lumbar radiculopathy . (Nervous system disorders) | 1 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Shoulder operation (Surgical and medical procedures) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aramchol 600mg (N=98) | Aramchol 400mg (N=101) | Placebo (N=48)
Abdominal distension (Gastrointestinal disorders) | 6 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 1
Asthenia (General disorders) | 5 | 4 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 1
Bronchitis (Infections and infestations) | 6 | 5 | 0
Constipation (Gastrointestinal disorders) | 8 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 4
Diarrhea (Gastrointestinal disorders) | 6 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 1
Fatigue (General disorders) | 3 | 8 | 4
Headache (Nervous system disorders) | 15 | 14 | 6
Influenza (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0
Nausea (Gastrointestinal disorders) | 9 | 10 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 7 | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
Urinary tract infection (Renal and urinary disorders) | 13 | 15 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consistent with scientific standards, publication of the results of the study shall be made only as part of a publication of the results obtained by all sites performing the protocol.

Investigators who wish to publish the results, must provide Galmed with a manuscript for review 60 (sixty) days prior to submission for publication.

Galmed retains the right to delete confidential and proprietary information and to object suggested publication and/or its timing (at the Company's sole discretion).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02279524/Prot_SAP_000.pdf